CLINICAL TRIAL: NCT05989061
Title: PEEK Versus Titanium Customized Healing Abutments: Evaluation of Peri-implant Soft Tissues and Sulcus Fluid Bacterial Load
Brief Title: PEEK Versus Titanium Customized Healing Abutments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Samar El Desouki, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RecIM122219
Record Dates: First submitted 2023-07-21; First posted 2023-08-14 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Dental Implants
Keywords: Customized Healing Abutment; PEEK; Peri-implant soft tissue; Dental implants; Titanium; Esthetic Zone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEEK customized healing abutment. (Experimental): Group I (Customized PEEK Healing Abutment):
  13 patients will receive guided delayed implant and a customized PEEK healing abutment placed simultaneously with implant surgery
  Interventions: Device: PEEK customized healing abutment
- Titanium customized healing abutment. (Active Comparator): Group II (Customized Titanium Healing Abutment):
  13 patients will receive guided delayed implant and a customized titanium healing abutment placed simultaneously with implant surgery.
  Interventions: Device: Titanium customized healing abutment

INTERVENTIONS:
Device: PEEK customized healing abutment — Guided delayed implant and a customized PEEK healing abutment placed simultaneously with implant surgery
  Arms: PEEK customized healing abutment.
Device: Titanium customized healing abutment — Guided delayed implant and a customized Titanium healing abutment placed simultaneously with implant surgery
  Arms: Titanium customized healing abutment.

SUMMARY:
The study suggests that if the investigators used customized healing abutments synthesized from PEEK may have a favorable effect on peri-implant soft tissues regarding decreased plaque accumulation and healing stimulation compared to the customized conventional titanium healing abutments.

DETAILED DESCRIPTION:
Successful aesthetic implant therapy has several sequential goals such as prosthetically driven 3D implant placement. Implant placement must be done in the ideal position to support the restoration and the surrounding soft and hard tissues. The placement of a definitive restoration should also be in harmony with the adjacent natural teeth and surrounding soft tissue.

Guided implant surgery can provide precise, predictable, and safe implant placement. Computer-generated surgical guides vary in design according to the dental condition (edentulous or partially edentulous), type of support (tooth, mucosa, or bone), and the degree of limitation (non-limiting, partially-limiting, or completely limiting).

The use of healing abutments has the function which enables adequate healing of peri-implant soft tissue and promoting a good profile of peri-implant mucosa that allows an adequate emergence profile of the prostheses supported by the implant. They are available in different lengths and project through the soft tissue into the oral cavity.

Janakievski stated that prefabricated healing abutments are unable to support the supracrestal soft tissues because of their circular profile. Therefore, a custom healing abutment is preferred because it provides a replica of the definitive restoration of the patient's gingival architecture.

An evaluation of the use of customized healing abutments has been performed aiming to assess possible advantages associated with this treatment modality. This procedure allows to maintain the peri-implant tissue and improve aesthetics until crown delivery. CAD/CAM enables the fabrication of high-quality implant abutments from solid blocks of different materials.

The contours of the healing abutment are based on the contours of a provisionally designed definitive prosthesis. The healing abutment promotes tissue healing and obtains contours that are well-matched with the contours of the definitive prosthesis.

Currently healing abutments made of polymers such as polyetheretherketone (PEEK) which have been used in orthopedic surgery, are used in dentistry, because of aesthetic & biological reasons maintaining the health of peri-implant soft tissues during healing.

Polyetheretherketone (PEEK) healing abutments can be chosen instead of titanium healing abutments because of their superior properties such as biocompatibility, inert chemical properties, white color, and decreased liability for biofilm accumulation.

Research Question "May PEEK healing abutment have a favorable effect on peri-implant soft tissue that may be related to the superior biological properties of PEEK regarding both decreased biofilm accumulation& healing stimulation?"

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be systematically free from any disease as according to Cornell Medical Index-Health Questionnaire .
2. Both genders.
3. Age from 20-50 years.
4. Missing tooth in esthetic zone (Anterior/Premolar) to be restored with standard implant, with no need for additional bone and soft tissue augmentation procedures.
5. Implants primary stability ISQ ≥ 70 unites using the Osstell Mentor
6. BuccoLingual bone width ≥ 6 mm.
7. Mesio distal space ≥ 7 mm
8. Sound Mesial and distal neighboring teeth.
9. At least 6 natural teeth remaining in the same arch .
10. Mouth opening ≥ 30mm.
11. Enough keratinized mucosa.
12. Thick phenotype.

Exclusion Criteria:

1. Poor oral hygiene condition.
2. Pregnant and lactating females.
3. Smokers.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of peri-implant soft tissue changes | 1 month after implantation and 4 months after implantation (just before prosthetic procedures)
  Clinical evaluation of peri-implant soft tissue changes the Probing Depth (PD).
Clinical evaluation of peri-implant soft tissue changes | 1 month after implantation and 4 months after implantation (just before prosthetic procedures)
  Clinical evaluation of peri-implant soft tissue changes the Plaque Index (PI) score.
Clinical evaluation of peri-implant soft tissue changes | 1 month after implantation and 4 months after implantation (just before prosthetic procedures)
  Clinical evaluation of peri-implant soft tissue changes the Gingival Index (GI)score.
Clinical evaluation of peri-implant soft tissue changes | 1 month after implantation and 4 months after implantation (just before prosthetic procedures)
  Clinical evaluation of peri-implant soft tissue changes the Gingival Bleeding Time Index (GBTI).
Clinical evaluation of peri-implant soft tissue changes | 1 month after implantation and 4 months after implantation (just before prosthetic procedures)
  Clinical evaluation of peri-implant soft tissue changes the Width of keratinized tissue (WKT).

SECONDARY OUTCOMES:
Biochemical evaluation | 1 month after implantation and 4 months after implantation (just before prosthetic procedures)
  Biochemical evaluation of peri-implant sulcus fluid (PISF) total bacterial load.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E. Amr, Assoc Prof, Study Director — Ain Shams University
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Baltayan S, Pi-Anfruns J, Aghaloo T, Moy PK. The Predictive Value of Resonance Frequency Analysis Measurements in the Surgical Placement and Loading of Endosseous Implants. J Oral Maxillofac Surg. 2016 Jun;74(6):1145-52. doi: 10.1016/j.joms.2016.01.048. Epub 2016 Feb 1. PMID 26917203
- [Background] Beretta M, Poli PP, Pieriboni S, Tansella S, Manfredini M, Cicciu M, Maiorana C. Peri-Implant Soft Tissue Conditioning by Means of Customized Healing Abutment: A Randomized Controlled Clinical Trial. Materials (Basel). 2019 Sep 19;12(18):3041. doi: 10.3390/ma12183041. PMID 31546800
- [Background] Cakan U, Delilbasi C, Er S, Kivanc M. Is it safe to reuse dental implant healing abutments sterilized and serviced by dealers of dental implant manufacturers? An in vitro sterility analysis. Implant Dent. 2015 Apr;24(2):174-9. doi: 10.1097/ID.0000000000000198. PMID 25706262
- [Background] Chen ST, Buser D. Clinical and esthetic outcomes of implants placed in postextraction sites. Int J Oral Maxillofac Implants. 2009;24 Suppl:186-217. PMID 19885446
- [Background] Chen ST, Buser D. Esthetic outcomes following immediate and early implant placement in the anterior maxilla--a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:186-215. doi: 10.11607/jomi.2014suppl.g3.3. PMID 24660198
- [Background] Chew M, Tompkins G, Tawse-Smith A, Waddell JN, Ma S. Reusing Titanium Healing Abutments: Comparison of Two Decontamination Methods. Int J Prosthodont. 2018 November/December;31(6):613-618. doi: 10.11607/ijp.5881. Epub 2018 Jul 30. PMID 30339159
- [Background] Cochran DL, Nummikoski PV, Schoolfield JD, Jones AA, Oates TW. A prospective multicenter 5-year radiographic evaluation of crestal bone levels over time in 596 dental implants placed in 192 patients. J Periodontol. 2009 May;80(5):725-33. doi: 10.1902/jop.2009.080401. PMID 19405825
- [Background] de Almeida EO, Pellizzer EP, Goiatto MC, Margonar R, Rocha EP, Freitas AC Jr, Anchieta RB. Computer-guided surgery in implantology: review of basic concepts. J Craniofac Surg. 2010 Nov;21(6):1917-21. doi: 10.1097/SCS.0b013e3181f4b1a0. PMID 21119455
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Finelle G, Lee SJ. Guided Immediate Implant Placement with Wound Closure by Computer-Aided Design/Computer-Assisted Manufacture Sealing Socket Abutment: Case Report. Int J Oral Maxillofac Implants. 2017 Mar/Apr;32(2):e63-e67. doi: 10.11607/jomi.4770. PMID 28291855
- [Background] Jemt T. Measurements of tooth movements in relation to single-implant restorations during 16 years: a case report. Clin Implant Dent Relat Res. 2005;7(4):200-8. doi: 10.1111/j.1708-8208.2005.tb00065.x. PMID 16336911
- [Background] Joda T, Ferrari M, Braegger U. A digital approach for one-step formation of the supra-implant emergence profile with an individualized CAD/CAM healing abutment. J Prosthodont Res. 2016 Jul;60(3):220-3. doi: 10.1016/j.jpor.2016.01.005. Epub 2016 Feb 9. PMID 26868927
- [Background] Lang LA, Sierraalta M, Hoffensperger M, Wang RF. Evaluation of the precision of fit between the Procera custom abutment and various implant systems. Int J Oral Maxillofac Implants. 2003 Sep-Oct;18(5):652-8. PMID 14579952
- [Background] Margonar R, Queiroz TP, Luvizuto ER, Betoni-Junior W, Zocal EA. Mandibular rehabilitation using immediate implant loading after computer-guided surgery. J Craniofac Surg. 2012 Mar;23(2):e129-32. doi: 10.1097/SCS.0b013e31824cdb74. PMID 22446446
- [Background] Mehra M, Somohano T, Choi M. Mandibular fibular graft reconstruction with CAD/CAM technology: A clinical report and literature review. J Prosthet Dent. 2016 Jan;115(1):123-8. doi: 10.1016/j.prosdent.2015.05.012. Epub 2015 Sep 11. PMID 26372630
- [Background] Molina A, Sanz-Sanchez I, Martin C, Blanco J, Sanz M. The effect of one-time abutment placement on interproximal bone levels and peri-implant soft tissues: a prospective randomized clinical trial. Clin Oral Implants Res. 2017 Apr;28(4):443-452. doi: 10.1111/clr.12818. Epub 2016 Mar 25. PMID 27016157
- [Background] Akoglan M, Tatli U, Kurtoglu C, Salimov F, Kurkcu M. Effects of different loading protocols on the secondary stability and peri-implant bone density of the single implants in the posterior maxilla. Clin Implant Dent Relat Res. 2017 Aug;19(4):624-631. doi: 10.1111/cid.12492. Epub 2017 May 10. PMID 28493347
- [Background] Pow EH, McMillan AS. A modified implant healing abutment to optimize soft tissue contours: a case report. Implant Dent. 2004 Dec;13(4):297-300. doi: 10.1097/01.id.0000144510.66524.87. PMID 15591990
- [Background] Priest G. Virtual-designed and computer-milled implant abutments. J Oral Maxillofac Surg. 2005 Sep;63(9 Suppl 2):22-32. doi: 10.1016/j.joms.2005.05.158. PMID 16125013
- [Background] Proussaefs P. Immediate provisionalization with a CAD/CAM interim abutment and crown: a guided soft tissue healing technique. J Prosthet Dent. 2015 Feb;113(2):91-5. doi: 10.1016/j.prosdent.2014.09.003. Epub 2014 Oct 28. PMID 25438739
- [Background] Pyo SW, Lim YJ, Koo KT, Lee J. Methods Used to Assess the 3D Accuracy of Dental Implant Positions in Computer-Guided Implant Placement: A Review. J Clin Med. 2019 Jan 7;8(1):54. doi: 10.3390/jcm8010054. PMID 30621034
- [Background] Rea M, Ricci S, Ghensi P, Lang NP, Botticelli D, Soldini C. Marginal healing using Polyetheretherketone as healing abutments: an experimental study in dogs. Clin Oral Implants Res. 2017 Jul;28(7):e46-e50. doi: 10.1111/clr.12854. Epub 2016 Apr 15. PMID 27080305
- [Background] Susin C, Finger Stadler A, Fiorini T, de Sousa Rabelo M, Ramos UD, Schupbach P. Safety and efficacy of a novel anodized abutment on soft tissue healing in Yucatan mini-pigs. Clin Implant Dent Relat Res. 2019 Mar;21 Suppl 1:34-43. doi: 10.1111/cid.12755. Epub 2019 Mar 12. PMID 30859699
- [Background] Wadhwani C, Schonnenbaum TR, Audia F, Chung KH. In-Vitro Study of the Contamination Remaining on Used Healing Abutments after Cleaning and Sterilizing in Dental Practice. Clin Implant Dent Relat Res. 2016 Dec;18(6):1069-1074. doi: 10.1111/cid.12385. Epub 2015 Dec 7. PMID 26640198
- [Background] Yunus N, Masood M, Saub R, Al-Hashedi AA, Taiyeb Ali TB, Thomason JM. Impact of mandibular implant prostheses on the oral health-related quality of life in partially and completely edentulous patients. Clin Oral Implants Res. 2016 Jul;27(7):904-9. doi: 10.1111/clr.12657. Epub 2015 Jul 14. PMID 26173463

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT05989061/Prot_SAP_000.pdf